CLINICAL TRIAL: NCT03281187
Title: A Randomized, Parallel, Double-dummy, Multi-center Phase III Study for Evaluation of Efficacy and Safety of Nasotestt Compared to Androgel Treating Hypogonadism in Male Research Participants.
Brief Title: Efficacy and Safety of Testosterone Nasal Gel for Treating Hypogonadism in Men.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: FBM Industria Brasileira Ltda (Industry)
Collaborators: Azidus Brasil Scientific Research and Development Ltda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TESFBM0717NA-III
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Hypogonadism
Keywords: Hormonal reposition, Testosterone nasal, Nasotestt
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Due to the differences on test and comparator product a double-dummy design will be used retaining the blind of the study. Therefore each participant will receive an active product and inactive medication (placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Nasotestt 5 mg (Experimental): Participants randomized to this arm must administer one packet of Nasotestt 5 mg in each nostril (3 times a day - T.I.D) for 60 days.
  Interventions: Drug: Nasotestt 5 mg; Other: Androgel Placebo
- Androgel 50 mg (Active Comparator): Participants randomized to this arm must administer one packet of Androgel 50 mg applied once daily to skin of shoulder for 60 days.
  Interventions: Drug: Androgel 50 mg; Other: Nasotestt Placebo
- Androgel Placebo (Placebo Comparator): Participants must administer one packet of Androgel placebo applied once daily to skin of shoulder in addition to an experimental drug for 60 days.
  Interventions: Drug: Nasotestt 5 mg; Other: Androgel Placebo
- Nasotestt Placebo (Placebo Comparator): Participants must administer one packet of Nasotestt Placebo in each nostril (3 times a day - T.I.D) in addition to an experimental drug for 60 days.
  Interventions: Drug: Androgel 50 mg; Other: Nasotestt Placebo

INTERVENTIONS:
Drug: Nasotestt 5 mg — The 114 participants randomized to this arm must administer one packet of testosterone 5 mg nasal gel (Nasotestt) in each nostril 3 times a day for 60 days.
  Other Names: Test Group
  Arms: Androgel Placebo; Nasotestt 5 mg
Drug: Androgel 50 mg — The 114 participants randomized to this arm must administer one packet of testosterone 50 mg topic gel (Androgel) applied once daily to skin of shoulders for 60 days.
  Other Names: Active Comparator Group
  Arms: Androgel 50 mg; Nasotestt Placebo
Other: Nasotestt Placebo — The participants randomized to this arm must administer one packet of placebo testosterone nasal gel (Nasotestt Placebo) in each nostril 3 times a day in addition to an active drug for 60 days.
  Other Names: Placebo Test Group
  Arms: Androgel 50 mg; Nasotestt Placebo
Other: Androgel Placebo — The participants randomized to this arm must administer one packet of placebo testosterone topic gel (Androgel Placebo) applied once daily to skin of shoulders in addition to an active drug for 60 days.
  Other Names: Placebo Comparator Group
  Arms: Androgel Placebo; Nasotestt 5 mg

SUMMARY:
This is a phase III study for evaluation of Nasotestt efficacy compared to Androgel in the treatment of male participants with hypogonadism condition (reduced levels of testosterone) that have clinical indication of hormonal replacement with testosterone.

DETAILED DESCRIPTION:
This efficacy and safety study will evaluate the superiority of Nasotestt (nasal gel) treatment compared to Androgel (topic gel) after 60 days of starting use. The efficacy endpoint will be verified through the percentage of participants which presented at the end of 60 days normalized levels of total testosterone (<300 ng/dL to >1050 ng/dL). Secondary efficacy endpoints will be collected throughout the study through: evaluation of symptoms of erectile dysfunction (The International Index of Erectile Function - IIEF), symptoms of prostatic disease (International Prostate Symptom Score - IPSS), measurement of abdominal perimeter and clinical global response to treatment (CGI-I questionnaire). As exploratory investigation, the satisfaction/comfort of Nasotestt use will be assessed by a specific questionnaire that will be applied to participants at the end of study. Safety evaluation data will include report of all adverse events, including type, frequency, intensity, seriousness, severity and action taken related to the investigational product of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male research participant, aged 18 years or older, with BMI between 18.50 and 32.00 kg/m2;
2. To present symptomatic or asymptomatic hypogonadism and serum total morning testosterone levels ≤ 300 ng / dL;
3. Laboratory evaluation of prostate specific antigen (PSA) levels within the normal range established by the laboratory or with non clinically significant changes (NCS) judged by the study Investigator;
4. Rhinoscopy and Glatzel mirror test normal or with changes that do not interfere with nasal absorption of medication Test;
5. Present healthy skin in the region of Comparator product application (skin of the shoulder).

Exclusion Criteria:

1. Diagnostic of prostatic and/or breast neoplasia;
2. PSA levels 4 ng/mL or higher, or 3 ng/mL or higher with elevated risk for prostatic neoplasia development;
3. Treatment with estrogens, gonadotropin releasing hormone (GnRH), growth hormone (GH) in the last 12 months;
4. Treatment with testosterone or any other androgen in the last two weeks (oral, buccal and topic), four weeks (intramuscular) or twelve weeks (implant) that precede randomization in the study;
5. Active rhinitis: allergic, seasonal, medicinal, vasomotor and atrophic;
6. Presence of grade II or III septum deviation (in any region of the nasal septum) and / or presence of nasal polyps or other conditions that determine nasal obstruction;
7. Hypersensibility of testosterone as well as to components present in the formulation of drugs.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2018-07-16 (Estimated); Primary Completion 2018-11-12 (Estimated); Study Completion 2020-01-13 (Estimated)

PRIMARY OUTCOMES:
Superiority Efficacy of Nasotestt comparing to Androgel on normalization of the blood testosterone levels | 60 days
  The success of treatment will be evaluated through statistical comparison of percentage of participants that achieved normal blood testosterone levels after 60 days of use.

SECONDARY OUTCOMES:
Improvement of erectile dysfunction symptoms | 60 and 90 days after starting treatment.
  Will be evaluated by statistical comparison between IIEF baseline values and results observed throughout study.
Improvement of prostatic symptoms | 60 and 90 days after starting treatment.
  Will be evaluated by statistical comparison between I-PSS baseline values and results observed throughout study.
Improvement of abdominal perimeter | 60 and 90 days after starting treatment.
  Will be evaluated by statistical comparison between baseline perimeter observed and other results obtained throughout study.
Global Clinical Response to treatment | 90 days after starting treatment.
  Will be assessed by a CGI - I questionnaire applied at the end of study. This instrument evaluate the improvement observed by physician throughout the study compared to condition observed at the baseline visit.
Incidence of adverse events | During 120 days
  Will be evaluated by periodic monitoring of adverse events, including changes in clinical laboratory parameters and vital signs occurred throughout the study.

OTHER OUTCOMES:
Satisfaction and comfort of Nasotestt use | After 120 days
  Will be evaluated by specific questionnaire application at the end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Silva, Director, Study Director — FBM Indústria Farmacêutica Ltda.

IPD SHARING:
Plan to Share IPD: Undecided
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data wil become public.